CLINICAL TRIAL: NCT03435224
Title: Desaturation Validation of INVSENSOR00012
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19088
Record Dates: First submitted 2018-02-05; First posted 2018-02-15 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00012 (Experimental): All subjects consented are enrolled into the test group and will receive the INVSENSOR00012.
  Interventions: Device: INVSENSOR00012

INTERVENTIONS:
Device: INVSENSOR00012 — Noninvasive pulse oximeter sensor

SUMMARY:
This study is designed to compare the accuracy of a noninvasive measurement of oxygen saturation compared to reference values obtained by a laboratory blood gas analyzer. Arterial blood samples will be collected from healthy adult subjects while undergoing a desaturation procedure wherein the concentration of oxygen inhaled is slowly reduced until the subject's arterial oxygen concentration is approximately 70%. During the desaturation, the subject's hand and arm without the arterial line will be subjected to motion.After completing the desaturation, the gas mixture will be returned to room air concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-50 years of age.
* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Hemoglobin value is greater than or equal to 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* Carbon monoxide (CO) value ≤ 2.0% fractional carboxyhemoglobin (FCOHb)
* Subject has a physical status of American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease (ASA I or II) as it applies to the systemic disease portion of the classification.
* Systolic Blood Pressure ≤ 140 mmHg and Diastolic Blood Pressure ≤ 90 mmHg.
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria:

* Subject is pregnant.
* Subject smokes (smoking includes e-cigarette use).
* Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has open wounds, inflamed tattoos or piercings, visible healing wounds.
* Subject experiences frequent or severe headaches and/or migraine headaches.
* Subject has known drug or alcohol abuse and/or use of recreational drugs.
* Subject has experienced a concussion or head injury with loss of consciousness within the last year.
* Subject has any chronic bleeding disorders (i.e. hemophilia).
* Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
* Subject has any cancer or history of cancer (not including skin cancer).
* Subject has a chronic neurological disease (i.e. multiple sclerosis, Huntington's Disease).
* Subject has any cardiac dysrhythmia(s) (i.e. atrial fibrillation) and has not received clearance by their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder) that interferes with the subject's level of consciousness.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator).
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject who has taken anticoagulant medication within the last 30 days.
* Subject has taken opioid pain medication within 24 hours of start of study.
* Subject has either signs or history of peripheral ischemia/carpal tunnel syndrome.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, plastic surgery, major ears, nose and throat (ENT) surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has donated blood within the past 30 days.
* Subject has symptoms of congestion, head colds, flu or other illnesses.
* Subject experiences claustrophobia or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
* Subject has chronic unresolved asthma, lung disease or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has heart conditions, insulin-dependent Diabetes or uncontrolled hypertension.
* Subject has given vaginal delivery, had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the last 6 months.
* Subject intends to participate in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours of the study.
* Discretion of investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 39 enrolled participants, 29 met inclusion criteria and proceeded to the study. The remainder of the enrolled participants include screen failures and subjects that did not proceed due to time constraints.
Period: Overall Study
Arm/Group | INVSENSOR00012
Started | 29
Completed | 25
Not Completed | 4
Not completed — Unable to achieve a minimum desaturation level | 4

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00012
Number analyzed (Participants) | 25
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0
  18-50 years | 25
  > 50 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 3
  Caucasian | 5
  Black or African American | 7
  Hispanic | 10

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation (SpO2) Accuracy of Sensor
Description: Performance of the sensors will be determined by comparing the noninvasive oxygen saturation measurement (SpO2) of the pulse oximeter sensors to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample and calculating the Arithmetic root mean square (ARMS) value.
Time Frame: 1-5 hours
Measure: Number; unit: % of oxygen saturated hemoglobin
Units Other Than Participants: blood samples
Arm/Group | INVSENSOR00012
Number analyzed (Participants) | 25
Number analyzed (blood samples) | 269
% of oxygen saturated hemoglobin | 1.99

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | INVSENSOR00012
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT03435224/Prot_SAP_000.pdf